CLINICAL TRIAL: NCT02950298
Title: Developmental Outcomes of School-aged Children With Infantile-onset Pompe Disease: A Telemedicine Approach to Assessment and Cognitive Training
Brief Title: Pompe Telemedicine Developmental Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00059526
Record Dates: First submitted 2016-06-22; First posted 2016-11-01 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Pompe Disease; Glycogen Storage Disease II
Keywords: Pompe; Glycogen Storage Disease II; Telemedicine; Duke University Medical Center
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The primary purpose of this study is to:

* Document the developmental outcomes of individuals with Pompe disease treated with long-term enzyme-replacement therapy (ERT) through school-age (ages 6-18) using measures of cognitive functioning, academic skills, and speech and language abilities.
* Investigate possible cognitive processing speed weaknesses using BrainBaseline neurocognitive assessment software.
* Investigate the relationship between behavior and other developmental factors including speech and language ability and cognitive ability.
* Explore if the use of selected iPad applications may help strengthen cognitive processing speed in children with Pompe disease

DETAILED DESCRIPTION:
The study will last approximately 2-3 years. It includes 2-4 visits to Duke for developmental assessments. The baseline/year 1 visit may take place at Duke (may take 1-2 days) or remotely via iPad. The follow up 1/year 2 visit may take place at Duke (1-2 days) or remotely via an iPad, depending upon each child's particular situation.

ELIGIBILITY:
Inclusion Criteria:

* Age range 6-18 years
* Diagnosis of classic Pompe disease by enzyme or molecular methods
* Patient, parent, or legal guardian is willing and able to give written informed consent
* English speaking child and care giver.

Exclusion Criteria:

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study is open to patients with classic Pompe disease.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-12; Primary Completion 2021-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Relationship between daily behaviors in school-aged children with Pompe disease and observed speech patterns, as assessed by speech pathology. | 2 years
Document the developmental outcomes and cognitive function of individuals with Pompe disease treated with long-term ERT through school-age (ages 6-18), as assessed by PPVT-4. | 2 years
  This outcome measure will be tested using measures testing cognitive function.
Document the developmental outcomes and language abilities of individuals with Pompe disease treated with long-term ERT through school-age (ages 6-18), as assessed by CELF-5. | 2 years
  This outcome measure will be tested using measures testing language abilities.
Document the developmental outcomes and cognitive function of individuals with Pompe disease treated with long-term ERT through school-age (ages 6-18), as assessed by Woodcock-Johnson Test of Achievement. | 2 years
Document the developmental outcomes and cognitive function of individuals with Pompe disease treated with long-term ERT through school-age (ages 6-18), as assessed by Leiter. | 2 years

SECONDARY OUTCOMES:
Relationship between daily behaviors in school-aged children with Pompe disease and development, as assessed by Conners. | 2 years
Relationship between daily behaviors in school-aged children with Pompe disease and development, as assessed by BRIEF-P. | 2 years
Relationship between daily behaviors in school-aged children with Pompe disease and development, as assessed by Child Behavior Checklist. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Mackey AP, Hill SS, Stone SI, Bunge SA. Differential effects of reasoning and speed training in children. Dev Sci. 2011 May;14(3):582-90. doi: 10.1111/j.1467-7687.2010.01005.x. Epub 2010 Nov 23. PMID 21477196
- [Background] Jones HN, Muller CW, Lin M, Banugaria SG, Case LE, Li JS, O'Grady G, Heller JH, Kishnani PS. Oropharyngeal dysphagia in infants and children with infantile Pompe disease. Dysphagia. 2010 Dec;25(4):277-83. doi: 10.1007/s00455-009-9252-x. Epub 2009 Sep 10. PMID 19763689
- [Background] Ebbink BJ, Aarsen FK, van Gelder CM, van den Hout JM, Weisglas-Kuperus N, Jaeken J, Lequin MH, Arts WF, van der Ploeg AT. Cognitive outcome of patients with classic infantile Pompe disease receiving enzyme therapy. Neurology. 2012 May 8;78(19):1512-8. doi: 10.1212/WNL.0b013e3182553c11. Epub 2012 Apr 25. PMID 22539577
- [Background] Kishnani PS, Steiner RD, Bali D, Berger K, Byrne BJ, Case LE, Crowley JF, Downs S, Howell RR, Kravitz RM, Mackey J, Marsden D, Martins AM, Millington DS, Nicolino M, O'Grady G, Patterson MC, Rapoport DM, Slonim A, Spencer CT, Tifft CJ, Watson MS. Pompe disease diagnosis and management guideline. Genet Med. 2006 May;8(5):267-88. doi: 10.1097/01.gim.0000218152.87434.f3. No abstract available. PMID 16702877